CLINICAL TRIAL: NCT05034536
Title: A Phase II Study of PD-1 Blockade With or Without LAG-3 Inhibition in Combination With Infliximab for the Treatment of Metastatic Melanoma and Prevention of Adverse Events
Brief Title: PD-1 Antibody Therapy + Infliximab for Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Ryan J Sullivan, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-077
Record Dates: First submitted 2021-08-29; First posted 2021-09-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Infliximab; relatlimab; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anti-PD-1 therapy + Infliximab (Experimental): Participants will be randomly assigned to receive physician's choice of anti-PD-1 therapy (pembrolizumab or nivolumab+relatlimab) and infliximab.
  * Pembrolizumab will be administered every 3 weeks for up to 2 years
  * Nivolumab+relatlimab will be administered every 4 weeks for up to 2 years
  * Infliximab will be administered on weeks 0, 2, and 6 (+/- 3 days) for a total of 3 doses
  Interventions: Drug: Pembrolizumab; Drug: Infliximab; Drug: Relatlimab; Drug: Nivolumab
- Anti-PD-1 therapy + Placebo (Experimental): Participants will be randomly assigned to receive physician's choice of anti-PD-1 therapy (pembrolizumab or nivolumab+relatlimab) and placebo.
  * Pembrolizumab will be administered every 3 weeks for up to 2 years
  * Nivolumab+relatlimab will be administered every 4 weeks for up to 2 years
  * Placebo. will be administered on weeks 0, 2, and 6 (+/- 3 days) for a total of 3 doses
  Interventions: Drug: Pembrolizumab; Drug: Placebo; Drug: Relatlimab; Drug: Nivolumab

INTERVENTIONS:
Drug: Pembrolizumab — Intravenous infusion
  Other Names: Keytruda
Drug: Infliximab — Intravenous infusion
  Other Names: AVSOLA; Ixifi; Remicade; Renflexis
  Arms: Anti-PD-1 therapy + Infliximab
Drug: Placebo — Intravenous infusion
  Arms: Anti-PD-1 therapy + Placebo
Drug: Relatlimab — Intravenous infusion
Drug: Nivolumab — Intravenous infusion

SUMMARY:
The purpose of this research is to test the safety and effectiveness of the investigational combination of anti-Programmed Death (PD)-1 antibody therapy with or without LAG-3 inhibition (pembrolizumab or nivolumab+relatlimab) and infliximab in treating metastatic melanoma.

DETAILED DESCRIPTION:
This is a randomized, double-blind, phase 2 clinical trial that combines anti-Programmed Death (PD)-1 antibody therapy with or without LAG-3 inhibition (pembrolizumab or nivolumab+relatlimab) with the anti-Tumor Necrosis Factor (TNF)-α antibody infliximab as first line treatment for the management of patients with metastatic or recurrent melanoma.

The U.S. Food and Drug Administration (FDA) has not approved infliximab for metastatic melanoma but it has been approved for other uses. The FDA has approved pembrolizumab as a treatment option for metastatic melanoma. The FDA has approved nivolumab+relatlimab as a treatment option for metastatic melanoma.

Pembrolizumab is a blocking antibody (a protein used in the immune system to identity and neutralize bacteria, viruses, and other foreign pathogens) that binds to PD-1 (a protein that helps regulate the immune system's response in the body) and blocks the interaction with PD-L1 and PD-L2 (proteins that inhibits the body's immune response). By blocking this interaction, it might lead to an anti-tumor immune response that may decrease tumor growth.

Relatlimab is believed to work by attaching to and blocking a molecule called Lymphocyte Activation Gene-3 (LAG-3). LAG-3 is a protein that is present on different types of cells in the immune system and controls parts of the immune system by shutting it down. Scientists believe that one way cancers escape the immune system is by shutting it down. Antibodies that block LAG-3 can potentially prevent LAG-3 from shutting down the immune system, thus allowing it to recognize and help the body destroy the cancer cells.

Nivolumab is believed to work by attaching to and blocking a molecule called PD-1. PD-1 is a protein that is present on different types of cells in the immune system and controls parts of the immune system by shutting it down. Antibodies that block PD-1 can potentially prevent PD-1 from shutting down the immune system, thus allowing it to recognize and help the body destroy the cancer cells.

Infliximab is an anti-TNFα agent (an antibody that blocks certain inflammatory hormones) that may interact with irEC (immune related (entero)colitis - inflammation that occurs in the digestive tract) which can develop among people with advanced melanoma. Anti- TNFα agents have shown to lead to rapid symptomatic improvement. By combining anti-PD-1 antibody therapy (pembrolizumab or nivolumab+relatlimab) and infliximab we believe it may lead to reduced immune related side effects while increasing effective anti-tumor immune response.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits. Participants will be randomized to receive either a) anti-PD-1 antibody therapy (pembrolizumab or nivolumab+relatlimab) plus infliximab or b) anti-PD-1 antibody therapy (pembrolizumab or nivolumab+relatlimab) plus placebo (an intravenous solution without medication). Participants will receive study treatment for as long as their disease does not worsen, they do not experience any unacceptable side effects, or they have completed the two years of anti-PD-1 antibody therapy. Participants will then be followed until the study doctor determines follow-up is no longer needed or until participant withdrawal. It is expected that about 36 people will take part in this research study A research grant, The Bridge Project, is supporting this research study by providing funding for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Participants must have histologically confirmed Stage III unresectable or Stage IV metastatic melanoma
* Patients should be treatment naïve and eligible for treatment with anti-PD-1 or anti-PD-1/LAG3 as a first line therapy (as selected by their treating physician)
* Patients previously treated for melanoma with surgical resection alone who present with recurrent Stage III unresectable or Stage IV metastatic melanoma are eligible for enrollment
* Patients who were previously treated with systemic neo-adjuvant or adjuvant anti-PD-1 therapy more than 6 months prior to study enrollment will be eligible. There are no restrictions to the use of prior BRAF targeted therapy.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan
* Diagnostic imaging studies such as MRIs and CT scans must be performed within 30 days of the date of registration
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes (WBC) > 3,000/uL
  * Absolute neutrophil count > 1,500uL
  * Platelets > 100,000/uL
  * Total bilirubin < 1.5 X institutional upper limits of normal; total bilirubin > 1.5X above institutional upper limits of normal will be allowed if direct bilirubin is within normal limits or if patients has a documented history of Gilbert's disease
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal and ≤5 ULN for patients with liver metastases
* Baseline laboratory measurements must be documented from tests within 14 days of the date of registration
* ECOG performance status ≤ 1 (see Appendix A)
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification which can be performed by the study investigators. To be eligible for this trial, participants should be class 2B or better
* Ability to understand and willingness to sign a written informed consent document
* Baseline tumor biopsies are required for all patients who have tumors that are deemed by the study investigators to be safely accessible

Exclusion Criteria:

* Patients with ocular or mucosal melanoma
* Participants previously treated with anti-PD1/PDL1/CTLA-4 monoclonal antibodies for metastatic or unresectable disease
* Patients who are receiving other anti-neoplastic agents
* Symptomatic or untreated leptomeningeal disease
* Patients carrying a diagnosis of immunodeficiency or receiving systemic steroid therapy (prednisone or equivalent > 10 mg/day) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Corticosteroids to prevent contrast reactions is allowable
* Patients with active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Prior history of inflammatory bowel disease, microscopic colitis or segmental colitis associated with diverticulosis
* Breastfeeding and pregnant women are excluded from this study since all anti-PD-1 drugs are class D agents with the potential for teratogenic or abortifacient effects.
* Uncontrolled intercurrent illness including, but not limited to:

  * A. Ongoing or active infection
  * B. Edema > Grade 1
  * C. Documented myocardial infarction or unstable/uncontrolled cardiac disease (eg, unstable angina, severe arrhythmias, congestive heart failure [New York Heart Association (NYHA) > Class II]) within 6 months of study entry
  * D. Arterial thrombosis or vascular ischemic events, such as transient ischemic attack, cerebral infarction, within 6 months prior to study entry
  * E. Serious or non-healing wound
  * F. History of any medical condition including cardiovascular disease or chronic obstructive pulmonary disease (COPD), that in the opinion of the investigator, may increase the risks associated with study participation or study treatments or may interfere with the conduct of the study or interpretation of study results
  * G. Psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
  * H. An elevated high-sensitivity troponin T level at baseline will be allowable as long as the patient has no evidence of active, clinically relevant cardiac disease.
* Patients with a history of a different malignancy are ineligible except for the following circumstances:

  * A. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy
  * B. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ and basal cell or squamous cell carcinoma of the skin
* Patients with a history of Hepatitis B infection (HBsAg reactive or HBCAB reactive) or Hepatitis C (HCV RNA is detected). Participants with a history of hepatitis C virus (HCV) infection may be enrolled if they have been treated and cured
* Patients with a history of latent or active granulomatous infection, including tuberculosis, histoplasmosis, or coccidiomycosis
* Has received a live vaccine within 30 days of planned start of study therapy
* Current bacterial infection requiring antibiotic treatment, or systemic fungal infection
* Patients with a known hypersensitivity to pembrolizumab, nivolumab, or relatlimab or any of its excipients
* Previous adverse reaction or hypersensitivity to infliximab
* Any prior immune-related adverse event while on adjuvant anti-PD-1-based immunotherapy with the following exceptions: any endocrine toxicity, any grade 1 or 2 toxicity that completely resolved; if there is uncertainty about the grade of prior toxicity, this will be adjudicated by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of immune-related adverse events (irAE) in patients treated with anti-PD-1 plus infliximab compared to pembrolizumab plus placebo | 12 weeks
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Incidence of severe immune-related adverse events (irAEs) (grade 3-5) in patients treated with anti-PD-1 antibody plus infliximab compared to anti-PD-1 antibody plus placebo | 12 weeks up to 2 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence of anti-PD-1 antibody cessation due to immune-related adverse events (irAEs) | 12 weeks up to 2 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence of clinically apparent infections in patients treated with anti-PD-1 antibody plus infliximab compared to anti-PD-1 antibody plus placebo | 12 weeks up to 2 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Overall survival rate of patients receiving combination anti-PD-1 antibody/infliximab compared with anti-PD-1 antibody/placebo | Time from randomization (or registration) to death due to any cause, or censored at date last known alive up to 2 years
  Analysis based on cumulative incidence, and will include competing risks of (a) steroid initiation, or (b) anti-PD-1 antibody cessation. The methods of Fine and Gray will be used for analysis.
Progression free survival rate of patients receiving combination anti-PD-1 antibody /infliximab compared with anti-PD-1 antibody/placebo | Time from randomization (or registration) to the earlier of progression or death due to any cause up to 2 years.
  Analysis based on cumulative incidence, and will include competing risks of (a) steroid initiation, or (b) anti-PD-1 antibody cessation. The methods of Fine and Gray will be used for analysis.
Response rate of patients receiving combination anti-PD-1 antibody/infliximab compared with anti-PD-1 antibody/placebo | Time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented up to 2 years
  Proportion of evaluable patients who achieve either a CR or PR per RECIST criteria
Cumulative steroid exposure (dose x duration) used for management of irAEs for anti-PD-1 antibody/infliximab compared to anti-PD-1 antibody/placebo patients | 12 weeks up to 2 years
  Calculated by adding the number of doses multiplied by strength of dose over the total follow-up time. Steroid exposure will be summarized descriptively for each treatment arm and compared using a Wilcoxon rank-sum test
Incidence of diarrhea in patients treated with anti-PD-1 antibody plus infliximab compared to anti-PD-1 antibody plus placebo | 12 weeks up to 2 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence of colitis in patients treated with anti-PD-1 antibody plus infliximab compared to anti-PD-1 antibody plus placebo | 12 weeks up to 2 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Sullivan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation